CLINICAL TRIAL: NCT02859363
Title: Improving the Diagnostic Rate of Fabry Disease in Patients With Cerebrovascular Involvement in Taiwan- a Cohort Screening Program
Brief Title: Fabry Disease in Cerebrovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Tsong-Hai Lee, Professor of Neurology, Chang Gung Memorial Hospital
Other Study IDs: Fabry Ver. 2_20160301_CGMH-LK
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young stroke: Historical DNA samples from projects 103-3254C (98-3889A3) and 100-4008C (97-0470B) will perform specific genetic testing for the 26 common Fabry mutation types in Taiwan.
  Interventions: Genetic: 26 common Fabry mutation types in Taiwan

INTERVENTIONS:
Genetic: 26 common Fabry mutation types in Taiwan — Historical DNA samples from projects 103-3254C (98-3889A3) and 100-4008C (97-0470B) will perform specific genetic testing.

SUMMARY:
Fabry disease is an X-linked disorder of glycosphingolipid catabolism caused by a deficiency of the enzyme α-galactosidase A (α-Gal A), which leads to a progressive accumulation of globotriaosylceramide (Gb-3) in plasma and tissue lysosomes throughout the body. Lysosomal accumulation can result in lysosomal and cellular dysfunction, which leads to renal, cardiac, and central nervous system (CNS) complications.

It is estimated that 1 in 40,000 males has Fabry disease, whereas the estimated prevalence in the general population is 1 in 117,000 people. Newborn screenings for both classical and atypical Fabry disease in Taiwan also revealed a markedly high incidence of 1 in 2,300 and 1 in 3,000 newborns. Cerebrovascular variant Fabry disease may affect up to 4.9% of male patients and 2.4% of female patients with idiopathic stroke.

The diagnosis of Fabry disease can be challenging due to the diverse signs and symptoms, different ages of onset, and variable timing and severity of progression. The importance of Fabry disease lies in the irreversible renal, cardiac, cerebrovascular, and neurological damage. An early diagnosis of Fabry disease is important for initiating symptom management and reducing life-threatening complications, as well as for early identification of other affected family members. Therefore, the present study would like to conduct further screening of high-risk group of early cerebrovascular involvement that is essential for the successful management of Fabry disease.

DETAILED DESCRIPTION:
This is a cross-sectional, population-based study to identify Fabry disease in patients with early cerebrovascular involvement. Eligible patients are age above 18 years old (<=55 years old) with early cerebrovascular involvement and have provided inform consent. Patients who have been diagnosed Fabry disease are not eligible.

The present study will use samples of early cerebrovascular involvement patients which have been enrolled in two previous IRB approved projects [103-3254C (origin 98-3889A3), 100-4008C (origin 97-0470B)], participants of both studies have consented that participants' samples could be further investigated if needed.

Since, the investigators cannot ensure whether the condition of enzyme activity of frozen plasma sample were decayed after long-term storage and the investigators don't have available normal range of enzyme activity of historical plasma sample, the investigators will perform specific genotyping of Fabry disease for these patients according to the specific mutation variants which have been identified in Taiwan population previously.

Patients will be recalled to assess Fabry related symptoms if genetic testing has mutation finding and family screening will be performed if applicable. Further inform consent will be obtained as well.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 y/o
* Both females and males who have ischemic or hemorrhagic stroke before the age of 55 y/o
* Patient or his/her legal representatives are willing to sign the informed consent

Exclusion Criteria:

* Ischemic or hemorrhagic stroke patients who are already diagnosed to have Fabry disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Historical DNA samples from projects 103-3254C (98-3889A3) and 100-4008C (97-0470B) will perform specific genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Conclusive diagnosis of Fabry disease | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke center, Department of Neurology, Linkou Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branton MH, Schiffmann R, Sabnis SG, Murray GJ, Quirk JM, Altarescu G, Goldfarb L, Brady RO, Balow JE, Austin Iii HA, Kopp JB. Natural history of Fabry renal disease: influence of alpha-galactosidase A activity and genetic mutations on clinical course. Medicine (Baltimore). 2002 Mar;81(2):122-38. doi: 10.1097/00005792-200203000-00003. No abstract available. PMID 11889412
- [Background] Kampmann C, Linhart A, Baehner F, Palecek T, Wiethoff CM, Miebach E, Whybra C, Gal A, Bultas J, Beck M. Onset and progression of the Anderson-Fabry disease related cardiomyopathy. Int J Cardiol. 2008 Nov 28;130(3):367-73. doi: 10.1016/j.ijcard.2008.03.007. Epub 2008 Jun 24. PMID 18572264
- [Background] Rolfs A, Bottcher T, Zschiesche M, Morris P, Winchester B, Bauer P, Walter U, Mix E, Lohr M, Harzer K, Strauss U, Pahnke J, Grossmann A, Benecke R. Prevalence of Fabry disease in patients with cryptogenic stroke: a prospective study. Lancet. 2005 Nov 19;366(9499):1794-6. doi: 10.1016/S0140-6736(05)67635-0. PMID 16298216
- [Background] Meikle PJ, Hopwood JJ, Clague AE, Carey WF. Prevalence of lysosomal storage disorders. JAMA. 1999 Jan 20;281(3):249-54. doi: 10.1001/jama.281.3.249. PMID 9918480
- [Background] Hwu WL, Chien YH, Lee NC, Chiang SC, Dobrovolny R, Huang AC, Yeh HY, Chao MC, Lin SJ, Kitagawa T, Desnick RJ, Hsu LW. Newborn screening for Fabry disease in Taiwan reveals a high incidence of the later-onset GLA mutation c.936+919G>A (IVS4+919G>A). Hum Mutat. 2009 Oct;30(10):1397-405. doi: 10.1002/humu.21074. PMID 19621417
- [Background] Liao HC, Chiang CC, Niu DM, Wang CH, Kao SM, Tsai FJ, Huang YH, Liu HC, Huang CK, Gao HJ, Yang CF, Chan MJ, Lin WD, Chen YJ. Detecting multiple lysosomal storage diseases by tandem mass spectrometry--a national newborn screening program in Taiwan. Clin Chim Acta. 2014 Apr 20;431:80-6. doi: 10.1016/j.cca.2014.01.030. Epub 2014 Feb 7. PMID 24513544
- [Background] Ries M, Ramaswami U, Parini R, Lindblad B, Whybra C, Willers I, Gal A, Beck M. The early clinical phenotype of Fabry disease: a study on 35 European children and adolescents. Eur J Pediatr. 2003 Nov;162(11):767-72. doi: 10.1007/s00431-003-1299-3. Epub 2003 Sep 20. PMID 14505049
- [Background] Mehta A, Ricci R, Widmer U, Dehout F, Garcia de Lorenzo A, Kampmann C, Linhart A, Sunder-Plassmann G, Ries M, Beck M. Fabry disease defined: baseline clinical manifestations of 366 patients in the Fabry Outcome Survey. Eur J Clin Invest. 2004 Mar;34(3):236-42. doi: 10.1111/j.1365-2362.2004.01309.x. PMID 15025684
- [Background] Lee SH, Li CF, Lin HY, Lin CH, Liu HC, Tsai SF, Niu DM. High-throughput detection of common sequence variations of Fabry disease in Taiwan using DNA mass spectrometry. Mol Genet Metab. 2014 Apr;111(4):507-12. doi: 10.1016/j.ymgme.2014.02.004. Epub 2014 Feb 17. PMID 24613481